CLINICAL TRIAL: NCT01713530
Title: A 26-week Trial Comparing Efficacy and Safety of Insulin Degludec/Insulin Aspart BID and Insulin Degludec OD Plus Insulin Aspart in Subjects With Type 2 Diabetes Mellitus Treated With Basal Insulin in Need of Treatment Intensification With Mealtime Insulin
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN5401-3996; 2012-002346-20 (EudraCT Number); U1111-1130-7135 (Other: WHO)
Record Dates: First submitted 2012-10-22; First posted 2012-10-24 (Estimated); Results first posted 2015-11-17 (Estimated); Last update posted 2018-04-02 (Actual); Status verified 2018-03

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — insulin degludec, insulin aspart drug combination; insulin degludec; Insulin Aspart

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- IDegAsp BID+/-OADs (Experimental)
  Interventions: Drug: insulin degludec/insulin aspart
- IDeg OD plus IAsp +/-OADs (Experimental)
  Interventions: Drug: insulin degludec; Drug: insulin aspart

INTERVENTIONS:
Drug: insulin degludec/insulin aspart — Dose individually adjusted. For subcutaneous (s.c, under the skin) administration twice a day.
  Arms: IDegAsp BID+/-OADs
Drug: insulin degludec — Dose individually adjusted. For subcutaneous (s.c, under the skin) administration once daily.
  Arms: IDeg OD plus IAsp +/-OADs
Drug: insulin aspart — Dose individually adjusted. For subcutaneous (s.c, under the skin) administration with the main meals 2-4 times daily in accordance with local labelling.
  Arms: IDeg OD plus IAsp +/-OADs

SUMMARY:
This trial is conducted in Africa, Europe and the United States of America (USA).

The aim of the trial is to compare the difference in change in glycosylated haemoglobin (HbA1c) between insulin degludec/insulin aspart (IDegAsp) and/or oral anti-diabetic drugs (OADs) and insulin degludec (IDeg) plus insulin aspart (IAsp)and/or OADs.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of type 2 Diabetes Mellitus at the discretion of the investigator for at least 26 weeks prior to screening (visit 1)
* Treatment with basal insulin for at least 12 weeks prior to randomisation with or without metformin, sulphonylurea (SU)/glinide, DPP-4 inhibitors, alfa-glucosidase-inhibitors
* HbA1c 7.0% - 10.0%
* Body mass index (BMI) less than or equal to 40.0 kg/m^2

Exclusion Criteria:

* Treatment with glucose-lowering agent(s) other than those stated in the inclusion criteria
* Stroke; heart failure New York Heart Association (NYHA) class III or IV; myocardial infarction; unstable angina pectoris; or coronary arterial bypass graft or angioplasty
* Chronic disorder or disease which might jeopardise safety or compliance
* Malignant neoplasms
* Recurrent severe hypoglycaemia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 274 (Actual)
Dates: Start 2013-02-21 (Actual); Primary Completion 2014-01-09 (Actual); Study Completion 2014-01-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (48):
- United States (25):
  - Novo Nordisk Investigational Site, Greenbrae, California
  - Novo Nordisk Investigational Site, Mission Hills, California
  - Novo Nordisk Investigational Site, San Diego, California
  - Novo Nordisk Investigational Site, Kissimmee, Florida
  - Novo Nordisk Investigational Site, Chicago, Illinois
  - Novo Nordisk Investigational Site, Indianapolis, Indiana
  - Novo Nordisk Investigational Site, Slidell, Louisiana
  - Novo Nordisk Investigational Site, Rockville, Maryland
  - Novo Nordisk Investigational Site, Buckley, Michigan
  - Novo Nordisk Investigational Site, Hillsborough, New Jersey
  - Novo Nordisk Investigational Site, Lawrenceville, New Jersey
  - Novo Nordisk Investigational Site, Toms River, New Jersey
  - Novo Nordisk Investigational Site, Greensboro, North Carolina
  - Novo Nordisk Investigational Site, Whiteville, North Carolina
  - Novo Nordisk Investigational Site, Kettering, Ohio
  - Novo Nordisk Investigational Site, Wadsworth, Ohio
  - Novo Nordisk Investigational Site, Pittsburgh, Pennsylvania
  - Novo Nordisk Investigational Site, Kingsport, Tennessee
  - Novo Nordisk Investigational Site, Austin, Texas
  - Novo Nordisk Investigational Site, Dallas, Texas
  - Novo Nordisk Investigational Site, Houston, Texas
  - Novo Nordisk Investigational Site, Round Rock, Texas
  - Novo Nordisk Investigational Site, San Antonio, Texas
  - Novo Nordisk Investigational Site, Tacoma, Washington
  - Novo Nordisk Investigational Site, Martinsburg, West Virginia
- Algeria (4):
  - Novo Nordisk Investigational Site, Algiers
  - Novo Nordisk Investigational Site, Annaba
  - Novo Nordisk Investigational Site, Constantine
  - Novo Nordisk Investigational Site, Oran
- Austria (6):
  - Novo Nordisk Investigational Site, Graz
  - Novo Nordisk Investigational Site, Innsbruck
  - Novo Nordisk Investigational Site, Linz
  - Novo Nordisk Investigational Site, Mödling
  - Novo Nordisk Investigational Site, Salzburg
  - Novo Nordisk Investigational Site, Vienna
- France (7):
  - Novo Nordisk Investigational Site, Caen
  - Novo Nordisk Investigational Site, La Roche-sur-Yon
  - Novo Nordisk Investigational Site, La Rochelle
  - Novo Nordisk Investigational Site, Le Creusot
  - Novo Nordisk Investigational Site, Montpellier
  - Novo Nordisk Investigational Site, Saint-Herblain
  - Novo Nordisk Investigational Site, Vénissieux
- Norway (6):
  - Novo Nordisk Investigational Site, Hamar
  - Novo Nordisk Investigational Site, Kongsvinger
  - Novo Nordisk Investigational Site, Kristiansand
  - Novo Nordisk Investigational Site, Oslo
  - Novo Nordisk Investigational Site, Skedsmokorset
  - Novo Nordisk Investigational Site, Stavanger

REFERENCES:
- [Result] Rodbard HW, Cariou B, Pieber TR, Endahl LA, Zacho J, Cooper JG. Treatment intensification with an insulin degludec (IDeg)/insulin aspart (IAsp) co-formulation twice daily compared with basal IDeg and prandial IAsp in type 2 diabetes: a randomized, controlled phase III trial. Diabetes Obes Metab. 2016 Mar;18(3):274-80. doi: 10.1111/dom.12609. Epub 2016 Jan 11. PMID 26592732
- [Result] Haluzik M, Fulcher G, Pieber TR, Bardtrum L, Tutkunkardas D, Rodbard HW. The co-formulation of insulin degludec and insulin aspart lowers fasting plasma glucose and rates of confirmed and nocturnal hypoglycaemia, independent of baseline glycated haemoglobin levels, disease duration or body mass index: A pooled meta-analysis of phase III studies in patients with type 2 diabetes. Diabetes Obes Metab. 2018 Jul;20(7):1585-1592. doi: 10.1111/dom.13261. Epub 2018 Mar 25. PMID 29451706
- [Derived] Yang W, Akhtar S, Franek E, Haluzik M, Hirose T, Kalyanam B, Kar S, Wu T, Gogas Yavuz D, Unnikrishnan AG. Postprandial Glucose Excursions in Asian Versus Non-Asian Patients with Type 2 Diabetes: A Post Hoc Analysis of Baseline Data from Phase 3 Randomised Controlled Trials of IDegAsp. Diabetes Ther. 2022 Feb;13(2):311-323. doi: 10.1007/s13300-021-01196-7. Epub 2022 Jan 19. PMID 35044568
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted in 5 countries (48 sites): Algeria (4), Austria (6), France (8), Norway (6) and United States (24).
Groups:
- IDegAsp BID: The subjects in this arm received insulin degludec/insulin aspart (IDegAsp) (100 U/mL, 3 mL prefilled pen PDS290) twice daily, subcutaneously in the abdomen, upper arm (deltoid area) or thigh either with breakfast and dinner or with lunch and dinner for 26 weeks. The subjects pre-study medication included a basal insulin regimen (insulin detemir; insulin glargine; insulin NPH) with or without oral anti-diabetic drugs (OADs) (metformin, sulphonylurea (SU), glinide, dipeptidyl peptidase-4 (DPP-4) inhibitors, α-glucosidase-inhibitors), for at least 12 weeks prior to visit 1 (screening).
- IDeg OD+IAsp: The subjects in this arm received IDeg (100 U/mL, 3 mL prefilled pen PDS290) once daily, subcutaneously in the abdomen, upper arm (deltoid area) or thigh at any time of the day. The subjects in this arm also received IAsp ([NovoRapid®/NovoLog®], 100 U/mL, 3 mL, FlexPen®) with the main meals 2-4 times daily, subcutaneously (preferably into the abdominal wall) in accordance with local labelling.
  The subjects pre-study medication included a basal insulin regimen (insulin detemir; insulin glargine; insulin NPH) with or without OADs (metformin, SU, glinide, DPP-4 inhibitors, α-glucosidase-inhibitors), for at least 12 weeks prior to visit 1.
Period: Overall Study
Arm/Group | IDegAsp BID | IDeg OD+IAsp
Started | 138 | 136
Exposed | 136 (One (1) subject was randomised in error and 1 subject withdrew consent) | 135 (One (1) subject was withdrawn by the investigator)
Completed | 113 | 117
Not Completed | 25 | 19
Not completed — Adverse Event | 0 | 5
Not completed — Withdrawal criteria | 21 | 12
Not completed — Unclassified | 4 | 2

BASELINE CHARACTERISTICS:
Population: The full analysis set (FAS) included all randomised subjects. The statistical evaluation of the FAS followed the intention-to-treat (ITT) principle and subjects contributed to the evaluation "as randomised".
Groups:
- Total: Total of all reporting groups
Arm/Group | IDegAsp BID | IDeg OD+IAsp | Total
Number analyzed (Participants) | 138 | 136 | 274
Age, Continuous [Mean (Standard Deviation); unit: years]
  Age | 59.6 (8.3) | 59.6 (9.2) | 59.6 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65 | 50 | 115
  Male | 73 | 86 | 159
Glycosylated haemoglobin (HbA1c) [Mean (Standard Deviation); unit: percentage of glycosylated haemoglobin] | 8.3 (0.9) | 8.3 (0.7) | 8.3 (0.8)
Fasting plasma glucose [Mean (Standard Deviation); unit: mmol/L] | 9.0 (3.0) | 8.8 (2.9) | 8.9 (3.0)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in HbA1c (%)
Description: Change from baseline in HbA1c (%) after 26 weeks of treatment
Time Frame: Week 0, week 26
Population: The FAS included all randomised subjects. The statistical evaluation of the FAS followed the ITT principle and subjects contributed to the evaluation "as randomised".
Measure: Least Squares Mean (Standard Error); unit: percentage change in HbA1c
Arm/Group | IDegAsp BID | IDeg OD+IAsp
Number analyzed (Participants) | 138 | 136
percentage change in HbA1c | -1.23 (0.13) | -1.42 (0.12)

2. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG)
Description: Change from baseline in FPG after 26 weeks of treatment
Time Frame: Week 0, week 26
Population: The FAS included all randomised subjects (2 subjects-baseline FPG not measured). The statistical evaluation of the FAS followed the ITT principle and subjects contributed to the evaluation "as randomised".
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | IDegAsp BID | IDeg OD+IAsp
Number analyzed (Participants) | 136 | 136
mmol/L | -2.22 (0.38) | -1.90 (0.36)

3. Secondary Outcome: Number of Treatment Emergent Hypoglycaemic Episodes
Description: According to the Novo Nordisk definition for confirmed hypoglycaemic episodes (severe hypoglycaemia and/or a measured Plasma Glucose (PG) <3.1 mmol/L(56 mg/dL))
Time Frame: During Weeks 0-26
Population: The safety Analysis Set (SAS): included all subjects who received at least one dose of the investigational product or its comparator. Subjects in the safety set contributed to the evaluation "as treated".
Measure: Number; unit: episodes
Arm/Group | IDegAsp BID | IDeg OD+IAsp
Number analyzed (Participants) | 136 | 135
episodes | 706 | 841

4. Secondary Outcome: Number of Treatment Emergent Hypoglycaemic Episodes
Description: According to the American Diabetes Association (ADA) definition following are the categories of hypoglycaemic episodes:
  Severe hypoglycaemia, Documented symptomatic hypoglycaemia, Asymptomatic hypoglycaemia, Probable symptomatic hypoglycaemia and Relative hypoglycaemia
Time Frame: During Weeks 0-26
Population: The SAS included all subjects who received at least one dose of the investigational product or its comparator. Subjects in the safety set contributed to the evaluation "as treated".
Measure: Number; unit: episodes
Arm/Group | IDegAsp BID | IDeg OD+IAsp
Number analyzed (Participants) | 136 | 135
episodes
  ADA (American Diabetes Association) | 2894 | 2685
  Severe | 29 | 15
  Documented symptomatic | 1818 | 1843
  Asymptomatic | 930 | 728
  Probable symptomatic | 26 | 33
  Relative | 91 | 66

5. Secondary Outcome: Number of Treatment Emergent Nocturnal (00:01-05:59 am) Confirmed Hypoglycaemic Episodes
Description: Nocturnal hypoglycaemic episodes are defined as occurring between 00:01 and 05:59 a.m.
Time Frame: Weeks 0-26
Population: as for outcome 4
Measure: Number; unit: episodes
Arm/Group | IDegAsp BID | IDeg OD+IAsp
Number analyzed (Participants) | 136 | 135
episodes | 75 | 96

6. Secondary Outcome: Incidence of Treatment Emergent Adverse Events (TEAE)
Description: A TEAE was defined as an event that has onset date on or after the first day of exposure to randomised treatment and no later than 7 days after the last day of randomised treatment
Time Frame: Weeks 0-26
Population: as for outcome 4
Measure: Number; unit: number of events
Arm/Group | IDegAsp BID | IDeg OD+IAsp
Number analyzed (Participants) | 136 | 135
number of events | 330 | 298

ADVERSE EVENTS:
Time Frame: The adverse events (AEs) were collected for a duration of 28 weeks ie. from the first trial-related activity after the subject had signed the informed consent until the end of the post-treatment follow-up period (visit 29).
Description: The SAS included all subjects who received at least one dose of the investigational product or its comparator. Subjects in the safety set contributed to the evaluation "as treated".
Arm/Group | IDegAsp BID | IDeg OD+IAsp
Serious Adverse Events (participants affected / at risk) | 7/136 | 13/135
Other Adverse Events (participants affected / at risk) | 46/136 | 38/135
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IDegAsp BID (N=136) | IDeg OD+IAsp (N=135)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0)
Atrioventricular block complete (Cardiac disorders) | 1 (1) | 0 (0)
Ocular hypertension (Eye disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 1 (1) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Wrong drug administered (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Hypersomnia (Nervous system disorders) | 1 (1) | 0 (0)
Hypoglycaemic unconsciousness (Nervous system disorders) | 1 (1) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1)
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Thrombosis (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IDegAsp BID (N=136) | IDeg OD+IAsp (N=135)
Diarrhoea (Gastrointestinal disorders) | 9 (9) | 9 (9)
Asthenia (General disorders) | 10 (10) | 2 (2)
Fatigue (General disorders) | 7 (7) | 1 (1)
Influenza (Infections and infestations) | 9 (9) | 5 (7)
Nasopharyngitis (Infections and infestations) | 11 (11) | 12 (14)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 7 (8)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8 (8) | 3 (3)
Headache (Nervous system disorders) | 10 (12) | 8 (12)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Novo Nordisk maintains the right to be informed of any Investigator plans for publication and to review any scientific paper, presentation, communication or other information concerning the investigation described in this protocol. Any such communication must be submitted in writing to the Novo Nordisk trial manager prior to submission for comments. Comments will be given within four weeks from receipt of the planned communication.